CLINICAL TRIAL: NCT03702842
Title: Transcutaneous Spinal Direct Current Stimulation to Enhance Locomotion After Spinal Cord Injury
Brief Title: Stimulation to Enhance Walking Post-SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Brooks Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201801582 -N -A; NIH/NICHD 5P2CHD08685 (Other Grant/Funding Number: REACT Center Pilot Studies Program); OCR16206 (Other: UF ID)
Record Dates: First submitted 2018-10-09; First posted 2018-10-11 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: SCI - Spinal Cord Injury; Incomplete Spinal Cord Injury
Keywords: walking; locomotor training; rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be randomized to receive either 16 sessions of locomotor training with lower or higher dosage tsDCS, but will be unaware of the stimulation dosage level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Immediate effects low dose tsDCS (Experimental): Participants will receive one session of walking with a lower dosage of stimulation using the Soterix Medical tsDCS stimulator. During each session, participants will be asked to walk for up to 30 minutes on a treadmill while the stimulation is delivered. Assessments will be completed before and after the bout of treadmill walking.
  Interventions: Device: Soterix Medical tsDCS stimulator; Other: Locomotor training
- Immediate effects higher dose tsDCS (Experimental): Participants will receive one session of walking with a higher dosage of stimulation using the Soterix Medical tsDCS stimulator. During each session, participants will be asked to walk for up to 30 minutes on a treadmill while the stimulation is delivered. Assessments will be completed before and after the bout of treadmill walking.
  Interventions: Device: Soterix Medical tsDCS stimulator; Other: Locomotor training
- Interventional effects: Lower dosage (Experimental): After completing the 2 sessions of the first part of the study, the participants will be randomized to two groups for the second part of the study. Those in the lower dosage group will receive 16 sessions of locomotor training with tsDCS stimulation applied at the lower dosage for up to 30 minutes using the Soterix Medical tsDCS stimulator. The training sessions will be scheduled 4 days per week for 4 weeks. All training will be overseen by a physical therapist with experience in SCI walking rehabilitation and will involve the use of an overhead support harness.
  Interventions: Device: Soterix Medical tsDCS stimulator; Other: Locomotor training
- Interventional effects: Higher dosage (Experimental): After completing the 2 sessions of the first part of the study, the participants will be randomized to two groups for the second part of the study. Those in the higher dosage group will receive 16 sessions of locomotor training with tsDCS stimulation applied at the higher dosage for up to 30 minutes using the Soterix Medical tsDCS stimulator. The training sessions will be scheduled 4 days per week for 4 weeks. All training will be overseen by a physical therapist with experience in SCI walking rehabilitation and will involve the use of an overhead support harness.
  Interventions: Device: Soterix Medical tsDCS stimulator; Other: Locomotor training

INTERVENTIONS:
Device: Soterix Medical tsDCS stimulator — tsDCS will be delivered to the lumbar region of the spinal cord with electrodes placed over the low back and abdomen. The electrodes will be secured with a large elastic bandage so that stimulation can be applied for up to 30 minutes during locomotor training with a harness attached to the ceiling for safety. A physical therapist will supervise the session.
Other: Locomotor training — Participants will complete 16 sessions of locomotor training (4 times per week for 4 weeks). This involves walking on a treadmill for up to 30 minutes with a harness attached to the ceiling for safety, followed by 10 minutes of overground walking training; with physical assistance as needed.

SUMMARY:
This pilot study will investigate the effects of transcutaneous direct current stimulation (tsDCS) on walking function in individuals with incomplete spinal cord injury. Following rehabilitation, individuals with ISCI often demonstrate improved walking function, but continue to have serious impairments that limit mobility, community participation and quality of life. Adjuvants to rehabilitation that increase spinal excitation during training may enhance its effectiveness. tsDCS is a non-invasive neuromodulation approach that uses a mild electrical current, applied over the skin of the low back, to alter the membrane potential of spinal neurons. tsDCS will be applied during locomotor training, a well-established rehabilitation strategy that promotes walking recovery. Locomotor training emphasizes repetitive and task-specific practice of coordinated walking, often with therapist assistance or cueing to promote high quality movement patterns. The study team will explore if tsDCS combined with locomotor training increases spinal excitation and thereby improves the effectiveness of walking rehabilitation.

DETAILED DESCRIPTION:
The purpose of this pilot study is to investigate the effects of transcutaneous direct current stimulation (tsDCS) on locomotor function and rehabilitation outcomes in individuals with incomplete spinal cord injury (ISCI). tsDCS is a mild, non-invasive form of electrical stimulation that can alter spinal cord excitability.

Specific Aim 1: To test the hypothesis that tsDCS applied during walking will improve motor activation in adults with chronic ISCI. A random order, double blind cross-over study will be conducted across two test sessions to compare the immediate effects of two dosages of tsDCS during walking. To assess motor activation, the primary outcome measure will be lower extremity surface electromyography.

Specific Aim 2 (Interventional): To test the hypothesis that tsDCS applied during 16 sessions of locomotor training will improve functional walking outcomes. Participants will be randomized to receive 16 sessions of locomotor training with one of the two tsDCS dosages. The primary outcome is walking function as measured by standardized clinical tests of walking speed and endurance.

To address the aims of the study, the investigators will use a two-part study design. Following phone and in-person screenings and physician approval, individuals will provide informed consent to the study procedures. In the first part, participants will complete two separate testing sessions, presented in random order, that involve up to 30 minutes of tsDCS at one of two dosages levels while walking. The researchers will assess changes in motor activation before and at the end of the period of walking. For the second part, participants will be randomized to receive 16 sessions of locomotor training with one of the two dosages of tsDCS. Before and after the 16-session intervention (i.e., at baseline and post intervention), the study team will assess functional outcomes through standardized tests of walking speed and endurance.

ELIGIBILITY:
Inclusion Criteria:

* Single spinal cord injury (duration >1 year) classified as neurologic level T12 or above based on the International Standards for the Neurologic Classification of Spinal Cord Injury, and classified on the American Spinal Cord Injury Association (ASIA) Impairment Scale (AIS) as 'C' or 'D' motor incomplete
* Capable of ambulating 10 feet with or without the use of gait devices, braces, or the assistance of one person
* Medically stable with no acute illness or infection
* Able to provide informed consent

Exclusion Criteria:

* Current diagnosis of an additional neurologic condition such as multiple sclerosis, Parkinson's disease, stroke, or brain injury
* Presence of unstable or uncontrolled medical conditions such as cardiovascular disease, myocardial infarction (<1 year), pulmonary infection or illness, renal disease, autonomic dysreflexia, infections, pain, heterotopic ossification
* Cognitive or communication impairments limiting communication with study staff or ability to provide informed consent
* Lower extremity joint contractures limiting the ability to stand upright and practice walking
* Skin lesions or wounds affecting participation in walking rehabilitation
* Acute or unstable fracture, diagnosis of osteoarthritis or bone impairments affecting safe participation in walking rehabilitation
* Severe spasticity or uncontrolled movements limiting participation in walking rehabilitation
* Body weight or height that is incompatible with safe use of a support harness and body weight support system
* Pain that limits walking or participation in walking rehabilitation
* Current participation in rehabilitation to address walking function
* Botox injections in lower extremity muscles affecting walking function within 4 months of study enrollment
* Legal blindness or severe visual impairment
* Known pregnancy
* Implanted metal hardware below the level of the 8th thoracic vertebrae

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2022-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emily Fox, PT, PhD, Principal Investigator — University of Florida
Locations (1):
- Brooks Rehabilitation Hospital, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled individuals were initially assigned to the 'Immediate effects' group. After completion of this arm, the same individuals were randomly assigned to either the Higher dosage or lower dosage interventional group (n=4 per group) Thus, only 8 individuals started and completed all procedures.
Groups:
- Part 1: Immediate Effects: tsDCS Lower Dose First, Then Higher Dose: lower dosage tsDCS using the Soterix Medical tsDCS stimulator followed by higher dosage tsDCS. During each session, participants will be asked to walk for up to 30 minutes on a treadmill while the stimulation is delivered. Assessments will be completed before and after the bout of treadmill walking.
  Soterix Medical tsDCS stimulator: tsDCS will be delivered to the lumbar region of the spinal cord with electrodes placed over the low back and abdomen. The electrodes will be secured with a large elastic bandage so that stimulation can be applied for up to 30 minutes during locomotor training with a harness attached to the ceiling for safety. A physical therapist will supervise the session.
  Soterix Medical tsDCS stimulator: tsDCS will be delivered to the lumbar region of the spinal cord with electrodes placed over the low back and abdomen. The electrodes will be secured with a large elastic bandage so that stimulation can be applied for up to 30 minutes during locomotor training with a harness attached to the ceiling for safety. A physical therapist will supervise the session.
- Part 2: Interventional Effects - Lower Dosage: After completing the 2 sessions of the first part of the study, the participants will be randomized to two groups for the second part of the study. Those in the lower dosage group will receive 16 sessions of locomotor training with tsDCS stimulation applied at the lower dosage for up to 30 minutes using the Soterix Medical tsDCS stimulator. The training sessions will be scheduled 4 days per week for 4 weeks. All training will be overseen by a physical therapist with experience in SCI walking rehabilitation and will involve the use of an overhead support harness.
  Soterix Medical tsDCS stimulator: tsDCS will be delivered to the lumbar region of the spinal cord with electrodes placed over the low back and abdomen. The electrodes will be secured with a large elastic bandage so that stimulation can be applied for up to 30 minutes during locomotor training with a harness attached to the ceiling for safety. A physical therapist will supervise the session.
  Locomotor training: Participants will complete 16 sessions of locomotor training (4 times per week for 4 weeks). This involves walking on a treadmill for up to 30 minutes with a harness attached to the ceiling for safety, followed by 10 minutes of overground walking training; with physical assistance as needed.
- Part 2: Interventional Effects - Higher Dosage: After completing the 2 sessions of the first part of the study, the participants will be randomized to two groups for the second part of the study. Those in the higher dosage group will receive 16 sessions of locomotor training with tsDCS stimulation applied at the higher dosage for up to 30 minutes using the Soterix Medical tsDCS stimulator. The training sessions will be scheduled 4 days per week for 4 weeks. All training will be overseen by a physical therapist with experience in SCI walking rehabilitation and will involve the use of an overhead support harness.
  Soterix Medical tsDCS stimulator: tsDCS will be delivered to the lumbar region of the spinal cord with electrodes placed over the low back and abdomen. The electrodes will be secured with a large elastic bandage so that stimulation can be applied for up to 30 minutes during locomotor training with a harness attached to the ceiling for safety. A physical therapist will supervise the session.
  Locomotor training: Participants will complete 16 sessions of locomotor training (4 times per week for 4 weeks). This involves walking on a treadmill for up to 30 minutes with a harness attached to the ceiling for safety, followed by 10 minutes of overground walking training; with physical assistance as needed.
Period: Part 1 Immediate Effects tsDCS Lower
Arm/Group | Part 1: Immediate Effects: tsDCS Lower Dose First, Then Higher Dose | Part 2: Interventional Effects - Lower Dosage | Part 2: Interventional Effects - Higher Dosage
Started | 8 | 0 | 0
Completed | 8 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part 1 Immediate Effects tsDCS Higher
Arm/Group | Part 1: Immediate Effects: tsDCS Lower Dose First, Then Higher Dose | Part 2: Interventional Effects - Lower Dosage | Part 2: Interventional Effects - Higher Dosage
Started | 8 | 0 | 0
Completed | 8 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Part 2 Interventional - Randomized
Arm/Group | Part 1: Immediate Effects: tsDCS Lower Dose First, Then Higher Dose | Part 2: Interventional Effects - Lower Dosage | Part 2: Interventional Effects - Higher Dosage
Started | 0 | 4 | 4
Completed | 0 | 4 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interventional Effects: Lower Dosage | Interventional Effects: Higher Dosage | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (12.3) | 53 (11.5) | 52 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 4 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 4 | 1 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in 10-Meter Walk Test (Interventional)
Description: Performance assessment of comfortable and fastest safe walking speed for 10 meters. A reduced time (in seconds) to complete the 10-Meter Walk Test reflects improvement in walking function.
Time Frame: Baseline; Week 4
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Interventional Effects: Higher Dosage | Interventional Effects: Lower Dosage
Number analyzed (Participants) | 4 | 4
meters/second | 0.18 (0.29) | -0.05 (0.23)

2. Primary Outcome: Change in Plantar Flexor Muscle Electromyogram Activation During Walking (Immediate Effects)
Description: The change in normalized amplitude of muscle activation recorded from the right ankle plantar flexor muscles (soleus and gastrocnemius) will be reported. EMGs will be recorded during speed-matched trials during walking on a treadmill. The normalized mean activation during single limb stance will be quantified for each step and averaged. For each participant, the change in activation will be quantified by subtracting activation pre training from post-training activation. The mean change and standard deviation of change will be reported for each group.
Time Frame: Baseline; 1 hour
Measure: Mean (Standard Deviation); unit: mV
Groups:
- Immediate Effects: Low Dose tsDCS: Participants will receive a single session of locomotor training with low dose tsDCS using the Soterix Medical tsDCS stimulator. During the session, participants will be asked to walk for up to 30 minutes on a treadmill while the stimulation is delivered. Assessments will be completed before and after the bout of treadmill walking.
  Soterix Medical tsDCS stimulator: tsDCS will be delivered to the lumbar region of the spinal cord with electrodes placed over the low back and abdomen. The electrodes will be secured with a large elastic bandage so that stimulation can be applied for up to 30 minutes during locomotor training with a harness attached to the ceiling for safety. A physical therapist will supervise the session.
- Immediate Effects: Higher Dose tsDCS: Participants will receive a single session of locomotor training with higher dose tsDCS using the Soterix Medical tsDCS stimulator. During the session, participants will be asked to walk for up to 30 minutes on a treadmill while the stimulation is delivered. Assessments will be completed before and after the bout of treadmill walking.
  Soterix Medical tsDCS stimulator: tsDCS will be delivered to the lumbar region of the spinal cord with electrodes placed over the low back and abdomen. The electrodes will be secured with a large elastic bandage so that stimulation can be applied for up to 30 minutes during locomotor training with a harness attached to the ceiling for safety. A physical therapist will supervise the session.
Arm/Group | Immediate Effects: Low Dose tsDCS | Immediate Effects: Higher Dose tsDCS
Number analyzed (Participants) | 8 | 8
mV | 0.0102 (0.1091) | -0.0023 (0.1257)

3. Secondary Outcome: Change in 6-Minute Walk Test (Interventional)
Description: The 6-Minute Walk Test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. An increase in the number of meters walked during this assessment reflects an improvement in walking endurance.
Time Frame: Baseline; Week 4
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Interventional Effects: Higher Dosage | Interventional Effects: Lower Dosage
Number analyzed (Participants) | 4 | 4
meters | 36.4 (69) | 4.9 (56.9)

ADVERSE EVENTS:
Time Frame: eight weeks
Description: Adverse events were collected in accordance with the definition used by clinicaltrials.gov. Additionally, participants were monitored during all study sessions using a standardized questionnaire and asked to report changes in health and function status.
Arm/Group | Part 1: Immediate Effects: tsDCS Lower Dose First, Then Higher Dose | Part 2: Interventional Effects - Higher Dosage | Part 2: Interventional Effects - Lower Dosage
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/8 | 3/4 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Immediate Effects: tsDCS Lower Dose First, Then Higher Dose (N=8) | Part 2: Interventional Effects - Higher Dosage (N=4) | Part 2: Interventional Effects - Lower Dosage (N=4)
skin abrasion or lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5) | 1 (1) — skin redness or abrasion
muscle tightness or spasm (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5) | 0 (0) — muscle spasticity or spasms
pain/discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-25): https://cdn.clinicaltrials.gov/large-docs/42/NCT03702842/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-04): https://cdn.clinicaltrials.gov/large-docs/42/NCT03702842/ICF_001.pdf